CLINICAL TRIAL: NCT01572103
Title: Coffee Consumption and Oxidative DNA Damage, Apoptosis and Collagen Synthesis in HCV-related Liver Disease: a Prospective Randomized Trial.
Brief Title: Coffee Effect in HCV-related Hepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Fabio Farinati, Associate Professor of Gastroenterology, Padua University, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ISIC
Record Dates: First submitted 2012-04-02; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Chronic HCV-related Hepatitis
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Administration of coffee (Experimental): Administration of 4 cups of coffee/day for 1 month
  Interventions: Dietary Supplement: Coffee
- Coffee abstinence (No Intervention): Total coffee and caffeine containing beverages abstinence
  Interventions: Dietary Supplement: coffee abstinence

INTERVENTIONS:
Dietary Supplement: Coffee — Administration of 4 cups of coffee per day for 1 month
  Arms: Administration of coffee
Dietary Supplement: coffee abstinence — total abstinence for both coffee and caffeine containing beverages
  Arms: Coffee abstinence

SUMMARY:
Background: In patients with chronic HCV-related liver damage, coffee is associated with a reduced risk of progression and of hepatocellular carcinoma (HCC) development. Aim: This prospective trial is aimed at assessing the mechanisms underlying the protective effect of coffee on evolution in cirrhosis and HCC. Trial design/methods: Forty patients with HCV-related hepatitis will be recruited and randomized into two groups: the first will consume 4 coffee cups/day/1 month, while the second will remain coffee "abstinent". At day 30, the two groups will be switched over and exposed to coffee or not for a second month. Before entering the study (time 0), during coffee exposure and during abstinence we will evaluate the following parameters: liver function tests, viral load, 8-hydroxydeoxyguanosine (a marker of oxidative DNA damage), telomere length, apoptosis and collagen deposition.

DETAILED DESCRIPTION:
Patients Forty patients with HCV-related chronic liver disease referring to the Gastroenterology Unit of Padua out-patient clinic will be prospectively recruited and will enter the study.

In all patients the presence of anti-HCV antibodies will be assayed by a third-generation immunoenzymatic test (Ortho Diagnostic Systems, Raritan, NJ) and by confirmatory test (recombinant immunoblotting assay, Chiron Corp., Emeryville, CA). A standardized genotyping assay (Inno-Lipa HCV III, Innogenetics, Gent, Belgium) will be used.

Only patients who fulfill the following inclusion criteria will be recruited:

* HCV-related chronic hepatitis or cirrhosis, with bioptic (within the previous 24 months) confirmation or a clinical diagnosis in case of cirrhosis; (Prothrombin Time - PT, White Blood Cells - WBC and platelets - PLT, Ultra Sound - US examination);
* anti-HCV and HCV-RNA positivity with Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) at least 1.5x;
* age range 30-80 years;
* no ongoing interferon treatment, previous treatment with no response or relapse was accepted.

The study is approved by the Hospital Ethical Committee (Prot. 1755 P, Azienda Ospedaliera di Padova), the patients' participation is voluntary and each patient signs an informed consent to participation, an information note being delivered to each patient's attending general practitioner.

Before the beginning of the intervention phase, for each patient, demographical data will be collected, together with information on coffee and smoking habits, alcohol, fruit, vegetable, anti-inflammatory drugs consumption, energy and nutrients intake, as potential bias. All these data will be assessed by using a quantity-frequency questionnaire designed for use in the present study. At time 0 (T0) the patients will be categorized into two groups in relation to their routine coffee intake: 0-2 cups/day and 3-5 cups/day. This cut-off was chosen because in most papers an effect of coffee consumption is observed for over 2 cups/day.

Subjects will be asked to maintain, throughout the study, their alimentary and voluptuary habits, while the use of other caffeine-containing beverages is forbidden.

Trial design of the study

Patients will be investigated for all the markers at the beginning of the study (T0) and then randomized using a computer-generated list (StatsDirect statistic program) in two groups, with either 4 coffee cups/day intake for 1 month or abstinence for the same time period. Obviously, blinding is not possible and we decided not to prescribe any wash-out period, being the T0 sampling examined in relation to the patients' routine coffee consumption.

After 30 days, the patients will be re-tested, and then shifted over to the opposite "treatment" (into the coffee arm those who were abstinent in the first month and vice versa those who consumed coffee) and again checked after the second time period.

Each patient is therefore tested three times, at T0, when he/she enters the study, after coffee and following abstinence, being each patient the control of himself in the two phases. For seek of simplicity all data obtained following coffee consumption will be compared with all the data obtained during abstinence, irrespective of the time sequence of exposure/abstinence.

Considering (on the basis of published data) an expected coffee effect in at least 40% of exposed subjects, with 1 control for case, with 5% alpha error and with 80% power, the sample size required (20 cases and 20 controls) corresponded to the selected sample for the study. Additionally, in this study, given the cross over design in which each patient is investigated twice, once during coffee exposure and once during abstinence, the actual number of patients investigated is of 40 per arm, twice as high therefore, than required.

The patients will be given a form in which they registered any deviation and compliance with respect to coffee intake and appropriate telephone contacts to report immediately any side effect. To reduce the risk of any bias due to inter-individual changes in the preparation of coffee, the patients will be provided with typical Italian-style coffee machine of the stove-top type (MokaTMBialetti), the required amount of coffee for the preparation of the 4 coffee cups/day (8 g for each coffee preparation) and instructions on how to prepare it.

The coffee brand is a 100% Coffea arabica product from the shelf. We also want to analyze the product we use. The analyses will be performed by a contract lab (Eurofins analytic GmbH - Hamburg-Germany).

The patients are instructed not to drink any differently prepared coffee and had to report in an appropriate form any deviation from the study.

Methods Blood samples will be collected and stored at -20°C for no longer than 3 weeks.

In this study the following parameters will be evaluated:

1. AST/ALT, gammaglutamyl-transpeptidase (γGT) and alkaline phosphatase (ALP) levels;
2. viral load (HCV-RNA titer),
3. markers of oxidative damage: 8-hydroxydeoxyguanosine (8-OHdG), nitric oxide (NO), Advanced Oxidation Protein Products (AOPP),
4. marker of genomic stability: Telomere Length (TL),
5. markers of cell death: M30 and M30/M65,
6. markers of liver fibrosis and angiogenesis: Procollagen Type III (PIIINP) and Vascular Endothelial Growth Factor (VEGF).

Liver Function Tests determination Serum levels of AST and ALT, gammaGT and ALP will be determined as part of the routine clinical procedure.

HCV-RNA determination The presence of HCV-RNA in the serum will be assessed by amplification with PCR of the 5' untranslated region (5'-UTR) of HCV, the most conserved region of the virus. The test is performed in all subjects positive for anti-HCV antibodies (screening test). The amplification will be performed in two steps, by 'nested PCR'.

8-OHdG determination This assay will be carried out as follows: in brief, this assay consists of 3 steps: (i) genomic DNA extraction using a Wizard Genomic DNA Purification Kit (Promega Italia, Milano); (ii) nuclease P1 and alkaline phosphatase hydrolysis of DNA; (iii) 8-OHdG determination using an HPLC equipped with an electrochemical detector (HPLC-ED) (ESA Coulochem II 5200 A, Bedford, MA). The 8-OHdG levels are expressed as the number of 8-OHdG adduct/105 dG.

NO determination Serum NO levels will be spectrophotometrically assayed by measuring the accumulation of its stable degradation products, nitrate and nitrite (Oxford Biomedical Research, USA). NO levels will be expressed as µmol/L, as a marker of nitric oxide synthase activation and nitrosation.

AOPP determination Plasma AOPP levels will be measured by spectrophotometric method performed by Witko-Sarsat. AOPP concentrations are expressed as µmol/L of chloramines-T equivalents.

TL analysis by quantitative PCR Genomic DNA extracted will be used also to measure TL by using method developed by Cawthon. Two 96-well plates were prepared for each experiment, one containing telomere primers and the other for 36B4, encoding acidic ribosomal phosphoprotein P0 used as the single copy gene .

Each 25 µl PCR reaction included 40 ng of DNA, SYBR Green Master Mix (Applied Biosystems, Foster City, CA) and primers at final concentrations 270 nM Tel-1 and 900 nM Tel-2 or 300 nM 36B4u and 500 nM 36B4d respectively.

PCR amplification is performed in a ABI PRISM 7900 (Applied Biosystem). In each plate, a standard curve is produced ranging from 4 to 80 ng of human reference DNA (Applied Biosystem). The thermal cycling profile for the telomere amplification is 95°C for 10 min, followed by 30 cycles of 95°C for 5 s, 56°C for 10 s and 72°C for 60 s or 30 cycles of 95°C for 5 s, 58°C for 10 s and 72°C for 40 s. Following amplification, a dissociation curve is performed in order to confirm the specificity of the reaction. All samples are assayed in triplicate to test the reproducibility of assay and in each assay a negative control is evaluated.

Fluorescence signals and dissociation curves are analyzed by ABI 7900 SDS 2.3 software.

Cell death determination The M30-Apoptosense ELISA (Peviva, USA) is a one step in vitro immunoassay for the quantitative determination of the apoptosis-associated CK18Asp396 (M30) neo-epitope in plasma. The concentration of the antigen that quantifies ongoing apoptotic cell death, is expressed as U/L.

The M30-Apoptosense ELISA is used in combination with M65 ELISA (Peviva, USA), for the quantitative determination of total soluble CK18 released from dead cells (necrotic and apoptotic). The concentration of the antigen is expressed as U/L.

PIIINP and VEGF determination Plasma PIIINP levels will be determined using ELISA kit (USCN, China). PIIINP levels are expressed as ng/mL as a marker of tissue collagen deposition and fibrosis. Serum VEGF will be determined as a marker of neo-angiogenesis and tissue re-modeling using an ELISA kit (Bender MedSystems, Austria), data being expressed in ng/L.

Statistic Data will be analyzed using one-way ANOVA, paired t-test, Student's t-test for unpaired data, linear regression (SPSS, STATSDIRECT) with statistical significance set at p <0.05 (2-tailed). All comparison regarding coffee exposure and abstinence will be carried within patients and not within groups, using, as said, a pair data approach.

ELIGIBILITY:
Inclusion Criteria:

* HCV-related chronic hepatitis or cirrhosis, with bioptic (within the previous 24 months) confirmation or a clinical diagnosis in case of cirrhosis (Prothrombin Time - PT, White Blood Cells - WBC and platelets - PLT, Ultra Sound - US examination suggestive for cirrhosis);
* anti-HCV and HCV-RNA positivity with AST/ALT at least 1.5x;
* age range 30-80 years;
* no ongoing interferon treatment, previous treatment with no response or relapse was accepted.

Exclusion Criteria:

* ongoing interferon treatment
* history of relevant cardiomyopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Variations in DNA oxidative damage levels following coffee exposure | Time0, 4 weeks and 8 weeks (exposure and abstinence, respectively)

SECONDARY OUTCOMES:
Effect of coffee exposure on changes in apoptosis | Time 0, 4 weeks and 8 weeks (exposure and abstinence, respectively)
Changes in collagen synthesis following coffee exposure in HCV-related hepatitis patients | Time 0, 4 weeks and 8 weeks (exposure and abstinence, respectively)